CLINICAL TRIAL: NCT02172014
Title: Safety and Efficacy of Fentanyl Citrate in Combination With Midazolam in Critically Ill Children With Mechanical Ventilation
Brief Title: Safety and Efficacy of Fentanyl Citrate in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, June Dong Park, MD, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MV_fentanyl
Record Dates: First submitted 2013-05-23; First posted 2014-06-24 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Children
Keywords: Mechanical Ventilation; Sedation; Fentanyl; Midazolam; Comfort behavior scale
MeSH Terms: interventions — Midazolam; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fentanyl (Experimental): midazolam and fentanyl citrate infusion
  Interventions: Drug: midazolam and fentanyl citrate infusion
- Control (Placebo Comparator): midazolam and normal saline infusion
  Interventions: Drug: midazolam and normal saline infusion

INTERVENTIONS:
Drug: midazolam and fentanyl citrate infusion — comparing the sedative effect of combination of midazolam and fentanyl citrate versus combination of midazolam and normal saline for 48 hours during ventilator care
  Other Names: midazolam injection; fentanyl citrate injection
  Arms: Fentanyl
Drug: midazolam and normal saline infusion — comparing the sedative effect of combination of midazolam and fentanyl citrate versus combination of midazolam and normal saline for 48 hours during ventilator care
  Other Names: midazolam injection
  Arms: Control

SUMMARY:
Title: Safety and efficacy of fentanyl citrate in combination with midazolam in critically ill children with mechanical ventilation

Objective: To evaluate the safety and efficacy of fentanyl citrate in combination with midazolam in children with mechanical ventilation.

Design: Double-blind randomized controlled study

Patients: Patients age 2 months through 18 years who are admitted in Seoul National University Hospital pediatric intensive care unit, and applied with mechanical ventilation.

Interventions: After enrollment of patient, blind reagent (fentanyl citrate or normal saline) is prepared by assigned pharmacist. Investigators, caregivers, patient, and parents of the patient don't know whether the blind reagent is fentanyl citrate or not, but only preparing pharmacist knows that.

Protocol: All enrolled patients receive continuous infusion of midazolam and blind reagent. The start time of study is when the continuous infusion of midazolam and blind reagent are begun. Assigned research nurse check Comfort behavior scale of the patient every hour regularly, and whenever the patient seem to be overactive. Endpoint of the study is 48 hours after begining. If there is any adverse effect or unexpected event, however, the study can be early terminated.

DETAILED DESCRIPTION:
Comfort behavior scale consists of 7 components of alertness, calmness, respiratory response, crying, physical movement, muscle tone, and facial tension. Because intubated patients cannot be evaluated 'crying', however, we use 6 components among total of all 7 components, except 'crying'.

Adverse effect of fentanyl include hypotension, coma, and ileus. Unexpected event means the situation which study cannot last in, such as withdrawal of consent, necessity of drugs which can affect the level of consciousness of the patient, emergent interventional procedure, etc.

ELIGIBILITY:
Inclusion Criteria:

* children mechanically ventilated
* age : from 2 months to 18 years

Exclusion Criteria:

* children with neurologic disease
* children with drugs which can affect the level of consciousness
* children with renal disease
* children with hypotension (systolic blood pressure < 70 + (2 x age in year) mmHg)

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2013-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
difference between measured Comfort behavior scale and target Comfort behavior scale | from the start of fentanyl/placebo infusion to 48 hours after start of infusion

SECONDARY OUTCOMES:
adverse effect | from the start of fentanyl/placebo infusion to 48 hour after start of infusion
  category of adverse effects
  1. hypotension
  2. coma
  3. ileus
renal dysfunction | from the start of fentanyl/placebo infusion to 48 hour after start of infusion
  estimate GFR (Schwartz equation) < 50 mL/minute/1.73m2
sedation failure | from the start of fentanyl/placebo infusion to 48 hour after start of infusion
  the case that can't reach target level of sedation, even though use of maximal infusion rate of midazolam and blind reagent.
mortality | from the start of fentanyl/placebo infusion to 48 hour after start of infusion
  in-hospital death

CONTACTS AND LOCATIONS:
Overall Officials: June Dong Park, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee B, Park JD, Choi YH, Han YJ, Suh DI. Efficacy and Safety of Fentanyl in Combination with Midazolam in Children on Mechanical Ventilation. J Korean Med Sci. 2019 Jan 7;34(3):e21. doi: 10.3346/jkms.2019.34.e21. eCollection 2019 Jan 21. PMID 30662387